CLINICAL TRIAL: NCT01929876
Title: A Phase 1, Open-Label Study to Evaluate the Effect of Itraconazole on the Pharmacokinetics of Cobimetinib in Healthy Subjects
Brief Title: A Study to Evaluate Effect of Itraconazole on the Pharmacokinetics of Cobimetinib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: GP28620
Record Dates: First submitted 2013-08-22; First posted 2013-08-28 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Participants
MeSH Terms: interventions — cobimetinib; Itraconazole

ARMS (1):
- Cobimetinib + Itraconazole (Experimental)
  Interventions: Drug: Cobimetinib; Drug: Itraconazole

INTERVENTIONS:
Drug: Cobimetinib — 10 milligram (mg) (2* 5 mg capsules) will be administered orally on Day 1 of Period 1 and Day 4 of Period 2
  Other Names: GDC-0973
Drug: Itraconazole — 200 mg oral solution will be administered once daily from Day 1 to Day 14 of Period 2

SUMMARY:
This open-label, 2-period, fixed sequence, drug interaction study will investigate the effect of co-administration of itraconazole on the pharmacokinetics of cobimetinib in healthy participants. Participants will receive multiple repeating doses of cobimetinib and itraconazole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult participants
* Within body mass index (BMI) range 18.5 to 32 kilogram per meter square (kg/m^2), inclusive
* Creatine phosphokinase levels below 2.5 times the upper limit of normal (ULN) and if elevated, not clinically significant
* Liver function tests for aspartate aminotransferase, alanine aminotransferase, and alkaline phosphatase below 2 times the ULN; bilirubin below 1.5 times the ULN; and all liver function test elevations not clinically significant
* In good health, determined by no clinically significant findings from medical history, 12-lead electrocardiogram (ECG), and vital signs
* Clinical laboratory evaluations within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator
* Negative test for selected drugs of abuse at screening and at each check-in
* Negative hepatitis panel (including hepatitis B surface antigen [HBsAg] and anti-hepatitis C virus [HCV]) and negative human immunodeficiency virus (HIV) antibody screens
* Females non-pregnant or non-lactating
* Males and females (of child-bearing potential) to use two forms of adequate contraception

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs; except that appendectomy, hernia repair, and/or cholecystectomy will be allowed
* History of diabetes mellitus and/or elevated fasting glucose at baseline
* History or presence of an abnormal ECG, which in the Investigator's opinion, is clinically significant
* History of alcoholism or drug addiction within 1 year prior to study start
* Use of any tobacco- or nicotine-containing products (within 6 months prior to study start and during the entire study
* Participation in any other investigational study or biologic agent trial in which receipt of an investigational study drug occurred within 5 half-lives or 30 days, whichever is longer, or exposure to any biological therapy or investigational biological agent within 90 days prior to study entry and during the entire study from study start to study completion, inclusive

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cobimetinib + Itraconazole: Cobimetinib 10 milligram (mg) (two 5 mg capsules) administered orally on Day 1 of Period 1 and Day 4 of Period 2. Each period duration was 14 days. Itraconazole 200 mg oral solution was administered once daily from Day 1 to Day 14 of Period 2.
Period: Period 1
Arm/Group | Cobimetinib + Itraconazole
Started | 16
Completed | 16
Not Completed | 0
Period: Period 2
Arm/Group | Cobimetinib + Itraconazole
Started | 16
Completed | 15
Not Completed | 1
Not completed — Non-Compliance | 1

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all participants who received at least 1 dose of cobimetinib and had at least 1 postdose safety assessment.
Groups:
- Cobimetinib + Itraconazole: Cobimetinib 10 mg administered orally on Day 1 of Period 1 and Day 4 of Period 2. Each period duration was 14 days. Itraconazole 200 mg oral solution was administered once daily from Day 1 to Day 14 of Period 2.
Arm/Group | Cobimetinib + Itraconazole
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Cobimetinib With and Without Itraconazole
Description: Maximum observed plasma concentration of cobimetinib with and without itraconazole was assessed using a model independent approach.
Time Frame: Period 1: Predose (0 hour), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 144, 192 hours postdose on Day 1; Period 2: Predose (0 hour), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 144, 192, 240 hours post cobimetinib dose on Day 4
Population: Pharmacokinetic (PK) population consisted of all participants who received at least 1 dose of cobimetinib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cobimetinib + Itraconazole
Number analyzed (Participants) | 15
nanogram per milliliter (ng/mL)
  Period 1: Cobimetinib Alone | 5.21 (38.1)
  Period 2: Cobimetinib With Itraconazole | 16.5 (27.7)
Statistical Analysis 1: Comparison: Cobimetinib + Itraconazole; Ratio of Least squares (LS) means (Cobimetinib with Itraconazole/Cobimetinib alone) of natural log-transformed parameter (expressed as a percent); Test type: Superiority or Other; Ratio of least squares means = 316.6, 90% CI 2-sided [268.1 to 374.0] — LS means from analysis of variance (ANOVA), calculated by transforming the natural log means back to the linear scale (that is, geometric LS mean)

2. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - Inf)] of Cobimetinib With and Without Itraconazole
Description: AUC (0 - inf) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf). It is obtained from AUC (0 - t) plus AUC (t - inf) of cobimetinib with and without itraconazole, assessed using a model independent approach.
Time Frame: as for outcome 1
Population: PK population. "Number of Participants Analyzed" indicates participants evaluable for this outcome measure and "n" signifies participants evaluable for specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cobimetinib + Itraconazole
Number analyzed (Participants) | 14
ng*hr/mL
  Period 1: Cobimetinib Alone (n=14) | 241 (51.5)
  Period 2: Cobimetinib With Itraconazole (n=12) | 1596 (23.0)
Statistical Analysis 1: Comparison: Cobimetinib + Itraconazole; Only participants with PK parameter data from both Period 1 Day 1 and Period 2 Day 4 (n=11) were included for statistical analyses; Test type: Superiority or Other; Ratio of LS means = 672.3, 90% CI 2-sided [563.7 to 801.9] — Ratio of LS means (Cobimetinib with Itraconazole/Cobimetinib alone) of natural log-transformed parameter (expressed as a percent). LS means from ANOVA, calculated by transforming the natural log means back to the linear scale

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Cobimetinib With and Without Itraconazole
Description: Time to reach maximum observed plasma concentration of cobimetinib with and without itraconazole was assessed using a model independent approach.
Time Frame: as for outcome 1
Population: PK population
Measure: Median (Full Range); unit: hours
Arm/Group | Cobimetinib + Itraconazole
Number analyzed (Participants) | 15
hours
  Period1: Cobimetinib Alone | 2.00 [1.00 to 6.05]
  Period 2: Cobimetinib With Itraconazole | 4.00 [2.00 to 8.02]

4. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] of Cobimetinib With and Without Itraconazole
Description: AUC (0-t) = Area under the plasma concentration versus time curve from time zero (predose) to time of last quantifiable concentration (0-t) of cobimetinib with and without itraconazole was assessed. It was calculated using the linear trapezoidal rule for increasing concentrations and the logarithmic rule for decreasing concentrations using a model independent approach.
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Cobimetinib + Itraconazole
Number analyzed (Participants) | 15
nanogram*hour per milliliter (ng*hr/mL)
  Period 1: Cobimetinib Alone | 209 (49.4)
  Period 2: Cobimetinib With Itraconazole | 1220 (24.0)
Statistical Analysis 1: Comparison: Cobimetinib + Itraconazole; Test type: Superiority or Other; Ratio of LS means = 583.9, 90% CI 2-sided [488.2 to 698.2] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Plasma Half-Life (t1/2) of Cobimetinib With and Without Itraconazole
Description: Plasma half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cobimetinib + Itraconazole
Number analyzed (Participants) | 14
hours
  Period1: Cobimetinib Alone (n=14) | 58.6 [25.9 to 89.2]
  Period 2: Cobimetinib With Itraconazole (n=12) | 118 [83.1 to 170]

6. Secondary Outcome: Apparent Clearance (CL/F) of Cobimetinib With and Without Itraconazole
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated using a model independent approach.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | Cobimetinib + Itraconazole
Number analyzed (Participants) | 14
liter per hour (L/hr)
  Period1: Cobimetinib Alone (n=14) | 41.4 (51.5)
  Period 2: Cobimetinib With Itraconazole (n=12) | 6.27 (23.0)

7. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Cobimetinib With and Without Itraconazole
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction of drug absorbed.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | Cobimetinib + Itraconazole
Number analyzed (Participants) | 14
liter (L)
  Period1: Cobimetinib Alone (n=14) | 3233 (27.5)
  Period 2: Cobimetinib With Itraconazole (n=12) | 1065 (36.1)

8. Secondary Outcome: Cmax of Itraconazole and Hydroxy-Itraconazole
Description: Maximum observed plasma concentration of itraconazole and its metabolite hydroxy-itraconazole was assessed using a model independent approach.
Time Frame: Period 2: Predose (0 hour), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 144, 192, 240 hours post cobimetinib dose on Day 4
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cobimetinib + Itraconazole
Number analyzed (Participants) | 15
ng/mL
  Itraconazole | 1480 (42.6)
  Hydroxy-Itraconazole | 1243 (26.4)

9. Secondary Outcome: Tmax of Itraconazole and Hydroxy-Itraconazole
Description: Time to reach maximum observed plasma concentration of itraconazole and its metabolite hydroxy-itraconazole was assessed using a model independent approach.
Time Frame: Period 2: Predose (0 hour), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 144, 192, 240 hours post cobimetinib dose on Day 4
Population: PK population
Measure: Median (Full Range); unit: hours
Arm/Group | Cobimetinib + Itraconazole
Number analyzed (Participants) | 15
hours
  Itraconazole | 2.00 [1.00 to 24.0]
  Hydroxy-Itraconazole | 4.00 [2.00 to 6.00]

10. Secondary Outcome: Area Under the Curve From Time Zero to 24 Hours [AUC (0-24)] of Itraconazole and Hydroxy-Itraconazole
Description: AUC (0-24) = Area under the plasma concentration versus time curve from time zero (predose) to 24 hours postdose (0-24) of itraconazole and its metabolite hydroxy-itraconazole was assessed using a model independent approach.
Time Frame: Period 2: Predose (0 hour), 0.5, 1, 2, 4, 6, 8, 12, 24 hours post cobimetinib dose on Day 4
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cobimetinib + Itraconazole
Number analyzed (Participants) | 15
ng*hr/mL
  Itraconazole | 15607 (26.8)
  Hydroxy-Itraconazole | 23176 (23.2)

ADVERSE EVENTS:
Time Frame: approximately 2 months
Description: Safety population
Arm/Group | Cobimetinib + Itraconazole
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 6/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cobimetinib + Itraconazole (N=16)
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Rhinitis (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.